CLINICAL TRIAL: NCT06570772
Title: Parallel-Group Treatment, Double-Blind, 2-Arm to Investigate Comparative Efficacy Safety Immunogenicity Between Intravenous AVT16 and Entyvio® in Male and Female Subjects 18 to 80 Years Inclusive, Moderate to Severe Ulcerative Colitis
Brief Title: Study to Investigate Comparative Efficacy, Safety and Immunogenicity Between AVT16 and Entyvio
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has been terminated based on Sponsor decision. This decision is not related to any safety concerns associated with the investigational products. It is related to the fact that study will be not required for product dossier submission.
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT16-GL-C01
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVT16 (Experimental): Experimental Arm AVT16 300mg iv is the proposed biosimilar for Entyvio (vedolizumab)
  Interventions: Biological: AVT16
- Entyvio (Active Comparator): Entyvio (vedolizumab) 300mg iv is the proposed active comparator for AVT16
  Interventions: Biological: Vedolizumab

INTERVENTIONS:
Biological: AVT16 — AVT16 will be given as iv infusion at Wks 0, 2, 6, 14, 22, 30, 38 and 46
  Other Names: AVT16 proposed biosimilar to vedolizumab
  Arms: AVT16
Biological: Vedolizumab — Entyvio (vedolizumab) will be given as iv infusion at Wks 0, 2, 6, 14, 22, 30, 38 and 46
  Other Names: Entyvio
  Arms: Entyvio

SUMMARY:
The study has been designed as a randomised, parallel-group, double-blind, 2 arm study of the comparative efficacy, safety and immunogenicity of AVT16 and Entyvio in male and female subjects with moderate to severe active ulcerative colitis.

DETAILED DESCRIPTION:
The study will consist of a screening period, a treatment and assessment period and an End of Study visit. Eligibility for the study will be determined during a screening period. Subjects who meet the eligibility criteria will be randomised to either AVT16 or Entyvio.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Male and female subjects from 18 to 80 years of age
* Diagnosis of Ulcerative Colitis

Exclusion Criteria:

* Diagnosis of Crohn's colitis
* Extensive colonic resection
* Active or latent tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Clinical Response at week 6 | Week 6
  Change in Mayo Score/Disease Activity for Ulcerative Colitis. Scale 0-12, higher score - worse outcome

SECONDARY OUTCOMES:
Clinical Response at week 52 | Week 52
  Change in Mayo Score/Disease Activity for Ulcerative Colitis. Scale 0-12, higher score - worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Schurink, Study Director — Alvotech Swiss AG
Locations (100):
- Argentina (4):
  - Investigational Site 161704, Ciudad Autónoma de BuenosAires
  - Investigational Site 161702, Córdoba
  - Investigational Site 161701, Quilmes
  - Investigational Site 161705, San Miguel de Tucumán
- Bulgaria (9):
  - Investigational Site 160111, Burgas
  - Investigational Site 160102, Pleven
  - Investigational Site 160109, Rousse
  - Investigational Site 160101, Sliven
  - Investigational Site 160103, Sofia
  - Investigational Site 160105, Sofia
  - Investigational Site 160108, Sofia
  - Investigational Site 160107, Stara Zagora
  - Investigational Site 160106, Vratsa
- Croatia (6):
  - Investigational Site 160204, Bjelovar
  - Investigational Site 160202, Osijek
  - Investigational Site 160205, Rijeka
  - Investigational Site 160206, Slavonski Brod
  - Investigational Site 160202, Zagreb
  - Investigational Site 160207, Zagreb
- Georgia (6):
  - Investigational Site 160507, Batumi
  - Investigational Site 160501, Tbilisi
  - Investigational Site 160502, Tbilisi
  - Investigational Site 160503, Tbilisi
  - Investigational Site 160505, Tbilisi
  - Investigational Site 160506, Tbilisi
- Latvia (3):
  - Investigational Site 160802, Liepāja
  - Investigational Site 160801, Riga
  - Investigational Site 160803, Riga
- Poland (27):
  - Investigational Site 161025, Bydgoszcz
  - Investigational Site 161008, Chojnice
  - Investigational Site 161013, Grudziądz
  - Investigational Site 161029, Kielce
  - Investigational Site 161018, Knurów
  - Investigational Site 161035, Krakow
  - Investigational Site 1614011, Ksawerów
  - Investigational Site 161028, Kłodzko
  - Investigational Site 161037, Lodz
  - Investigational Site 161015, Lublin
  - Investigational Site 161033, Olsztyn
  - Investigational Site 161021, Piotrkow Trybunalski
  - Investigational Site 161022, Poznan
  - Investigational Site 161023, Rzeszów
  - Investigational Site 161024, Rzeszów
  - Investigational Site 161009, Sopot
  - Investigational Site 161014, Swidnica
  - Investigational Site 161010, Szczecin
  - Investigational Site 161005, Torun
  - Investigational Site 161017, Tychy
  - Investigational Site 161007, Warsaw
  - Investigational Site 161012, Warsaw
  - Investigational Site 161016, Warsaw
  - Investigational Site 161041, Warsaw
  - Investigational Site 161006, Wroclaw
  - Investigational Site 161040, Wroclaw
  - Investigational Site 161026, Zamość
- Romania (3):
  - Investigational Site 161102, Constanța
  - Investigational Site 161103, Târgu Mureş
  - Investigational Site 161101, Timișoara
- Serbia (10):
  - Investigational Site 161201, Belgrade
  - Investigational Site 161203, Belgrade
  - Investigational Site 161204, Belgrade
  - Investigational Site 161206, Belgrade
  - Investigational Site 161209, Belgrade
  - Investigational Site 161205, Leskovac
  - Investigational Site 161211, Niš
  - Investigational Site 161207, Novi Sad
  - Investigational Site 161202, Pančevo
  - Investigational Site 161208, Zrenjanin
- Slovakia (6):
  - Investigational Site 161304, Banská Bystrica
  - Investigational Site 161303, Bratislava
  - Investigational Site 161301, Košice
  - Investigational Site 161302, Prešov
  - Investigational Site 161305, Rimavská Sobota
  - Investigational Site 161306, Trnava
- Sri Lanka (5):
  - Investigational Site 162204, Colombo
  - Investigational Site 162203, Galle
  - Investigational Site 162206, Jaffna
  - Investigational Site 162205, Kandy
  - Investigational Site 162201, Ragama
- Ukraine (21):
  - Investigational Site 160411, Cherkasy
  - Investigational Site 160401, Chernivtsi
  - Investigational Site 160412, Ivano-Frankivsk
  - Investigational Site 160404, Kyiv
  - Investigational Site 160405, Kyiv
  - Investigational Site 160406, Kyiv
  - Investigational Site 160413, Kyiv
  - Investigational Site 160416, Kyiv
  - Investigational Site 160420, Kyiv
  - Investigational Site 160422, Kyiv
  - Investigational Site 160425, Kyiv
  - Investigational Site 160407, Lviv
  - Investigational Site 160409, Lviv
  - Investigational Site 160417, Lviv
  - Investigational Site 160408, Uzhhorod
  - Investigational Site 160403, Vinnytsia
  - Investigational Site 160410, Vinnytsia
  - Investigational Site 160415, Vinnytsia
  - Investigational Site 160421, Vinnytsia
  - Investigational Site 160424, Vinnytsia
  - Investigational Site 160419, Zhytomyr

IPD SHARING:
Plan to Share IPD: No